CLINICAL TRIAL: NCT04581863
Title: Randomized Trial of Adding Pulse Oximetry to an Automated Text-messaging Program for Remotely Monitoring Patients at Home With COVID-19
Brief Title: COVID-19 Watch + COVID-19 Pulse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 844043
Record Dates: First submitted 2020-10-07; First posted 2020-10-09 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- COVID Watch (Active Comparator): COVID Watch provides text-based assessments, two times a day for 14 days and escalates care to a nurse via telemedicine for any reported worsening of symptoms not severe enough to recommend going to the ED immediately. This service is provided free of charge to patients, a benefit to patients without insurance or established primary care. UPHS already offers a version of COVID Watch with pulse oximetry to patients with COVID-19 being discharged from the ED who meet specific criteria: a discharge pulse ox less than 95%, an infiltrate on chest x-ray, are or age of 60 years or older, or who are deemed by the ED clinician to have significant comorbid conditions.
  Interventions: Other: COVID Watch
- PCORI Pulse (Experimental): This arm is COVID Watch + pulse oximeter device. Patients sent a pulse oximeter will be prompted twice daily to text their oxygen saturation level after walking in place for 1 minute. If the oxygen saturation is >3% lower than than the baseline first O2 sat measurement, or if it falls below an absolute level of 90%, the patient will receive an immediate call from the same on-call RN's for COVID Watch and undergo the same triage protocol .
  Interventions: Device: pulse oximeter; Other: COVID Watch

INTERVENTIONS:
Device: pulse oximeter — Patients will be prompted twice daily to text their oxygen saturation level after walking in place for 1 minute. If the oxygen saturation is >3% lower than than the baseline first O2 sat measurement, or if it falls below an absolute level of 90%, the patient will receive an immediate call from the same on-call RN's for COVID Watch and undergo the same triage protocol .
  Arms: PCORI Pulse
Other: COVID Watch — Enrolled patients receive text-based assessments, two times a day for 14 days and escalates care to a nurse via telemedicine for any reported worsening of symptoms not severe enough to recommend going to the ED immediately.

SUMMARY:
The clinical guidance for 90 percent of infected COVID-19 adult patients who do not meet eligibility for inpatient admission is to self-isolate. To support these patients, alternatives to in-person care are needed to manage an unpredictable clinical course; identify and intercept patients rapidly deteriorating at home, prevent viral spread during in-person visits; and minimize future surges in emergency departments (EDs). In addition, fingertip pulse oximeters have been proposed to improve in-home early detection of respiratory deteriorations but are untested and the operational infrastructure to support large-scale monitoring is limited.

While telemedicine has been widely adopted during the pandemic as an alternative to conventional outpatient care, limited telemedicine access may be exacerbating observed disparities for Black and Latino patients. In our health system, Black and Latino patients used video-visits 15 percent less often than white patients. Text messaging and phone calls may improve healthcare access for communities of color, but the evidence for these telecommunication modalities to be effective and improve equity are limited.

The University of Pennsylvania Health System (UPHS) developed and deployed COVID Watch to improve access to health care for COVID-19 patients who are self-isolating at home. COVID Watch sends twice-daily, scheduled text messages to assess patients for shortness of breath using a clinical algorithm to determine whether patients need an urgent escalation to a team of dedicated, on-call nurses within one hour. These nurses are supported by an on-call team of clinicians who can conduct urgent phone or video assessments. Patients can also trigger the algorithmic assessment independent of the scheduled messages. As of May 21, 2020, COVID Watch has managed 3,628 COVID-19 patients at home, of which 1,295 are confirmed COVID-19 positive; of these, 61 percent are Black or Latino, higher than the proportion of all UPHS COVID-19 positive patients that are Black or Latino (55 percent).

DETAILED DESCRIPTION:
Most (80-90%) COVID-19 positive patients are asked to self-isolate at home because they do not qualify for home care or inpatient admission. Alternatives to in-person care are urgently needed to: (1) manage an unpredictable clinical course; (2) identify and intercept patients rapidly deteriorating at home, (3) prevent viral spread during in-person visits; and (4) triage symptoms to minimize surges to emergency departments (EDs). In addition, fingertip pulse oximeters ("pulse oximetry") have been proposed to improve in-home early detection of respiratory deteriorations but are untested and the operational infrastructure to support large-scale monitoring is limited. While telemedicine has been widely adopted during the pandemic as an alternative to conventional outpatient care, worse COVID-19 outcomes observed among Black and Latino patients may be due, in part, to worse telemedicine access for these socially and medically disadvantaged groups.

To improve in-home monitoring and health care access for patients with suspected or confirmed COVID-19, the health innovation team at University of Pennsylvania Health System ("UPHS") developed COVID Watch, a free of charge, 24/7, automated, text message-based, home monitoring program across UPHS' large geographic catchment area. This study will answer the question, "How does the addition of pulse oximetry affect clinical outcomes for COVID-19 patients?"

COVID Watch was first implemented on March 24, 2020 and has enrolled 3,628 patients through May 21, 2020 of which 1,295 were COVID-19 positive. Understanding the effect of COVID Watch with and without pulse oximetry on Black and Latino patients is important because communities of color have had disproportionately higher rates of COVID-19 morbidity and mortality nationally, and locally in Pennsylvania, ranking 5th total deaths, and New Jersey, ranking 2nd. Symptom monitoring apps and programs are commercially available. However, COVID Watch is uniquely embedded into its host healthcare system, UPHS. Patients are enrolled using the electronic medical record (EMR), escalations are addressed by UPHS nurses, and they are referred to UPHS-based telemedicine, primary care, and social services when appropriate. COVID Watch is a scalable operational platform for monitoring patients with home pulse oximetry readings. Whether remote monitoring with or without pulse oximetry helps COVID-19 patients stay safe at home is an urgent, patient-centered question. Finally, with COVID-19 surges projected in late 2020, health systems will need to be prepared with evidence-based strategies for managing more COVID-19 patients at home.

COVID Watch (https://covidwatch.waytohealth.org/) is powered by UPHS' NIH-funded research and operational texting platform (www.waytohealth.org), integrated with UPHS' EMR. Since hypoxemia is the primary driver of admission and fatality among COVID-19 patients, the investigators focused the algorithm on shortness of breath, our closest approximation for concerning hypoxemia. Given the rapid and unpredictable decompensation of COVID-19 patients, patients receive clinical support 24 hours/day, 7 days/week. COVID Watch sends twice-daily, scheduled text messages to assess patients for shortness of breath using an algorithm to determine whether patients need an urgent escalation to a team of dedicated nurses within 1 hour. These nurses are supported by an on-call team of clinicians who can conduct urgent phone or video assessments. At each level patients' clinical needs are either managed with self-care advice, prescriptions, or a referral to the ED. The majority of COVID Watch patients (83.7%) have been enrolled by outpatient providers conducting telephone and video visits; 8.7% and 7.6% have been enrolled at ED and inpatient discharge, respectively. The program is available at all six of UPHS's hospitals and EDs, and all 530 affiliated ambulatory settings using the EMR. Any clinical staff member (e.g., RN, physician, medical assistants) logged on to the EMR is able to enroll patients. Patients can also trigger the algorithmic assessment independent of the scheduled messages. Patients only continue the intervention if they are agreeable ("opt-out") and can stop anytime. Patients are scheduled to be in COVID Watch for 14 days, with the option to extend to 21 days if interested. A Spanish-language version of COVID Watch was made available to patients on May 18, 2020, with nurses using translation lines to communicate with patients.

COVID Watch engagement is high. To date, nearly 80% of enrolled patients have engaged with the program, defined as responding to scheduled text messages at least once every two days. RNs have managed over 600 calls with a mean response time (median) of 25 minutes (11 minutes). Of the calls, 37% were asked to continue to monitor at home, 41% were scheduled for an urgent follow-up telemedicine visit, and 9% were sent to the ED for emergent evaluation.

The investigative team provides a conceptual model of how adding home pulse oximetry may potentially improve outcomes. Preventing or aggressively treating respiratory failure is essential for patients infected with COVID-19. Among all infected patients, an estimated 10-20% of patients with COVID-19 develop severe illness requiring hospitalization, of which 30-40% develop critical illness requiring support in an intensive care unit. Among the critically ill, respiratory failure is common and results from acute hypoxemic respiratory failure due to acute respiratory distress syndrome (ARDS). ARDS is a clinical manifestation of pulmonary tissue inflammation, preventing the exchange of oxygen between inhaled air and blood circulating in patients' lungs ("hypoxemia"). Increasing the concentration of oxygen in the air that patients breathe (e.g., supplemental oxygen) and reducing the degree of pulmonary inflammation can support patients with COVID-19 by reducing the severity of hypoxemia and providing sufficient oxygen supply to vital organs. Measures of pulse oximetry - the oxygen saturation in the blood - can provide an objective measure to identify which patients have or are beginning to experience declines in their respiratory function.

The investigators' conceptual model is based on emerging evidence that early medical interventions can improve clinical outcomes for COVID-19, resulting in less severe clinical sequelae and reduced mortality. For COVID-19 patients requiring supplemental oxygen, new preliminary data from a large multicenter randomized controlled trial of dexamethasone indicates that patients have markedly reduced mortality when given dexamethasone. This corticosteroid likely reduces pulmonary inflammation and prevents the development of severe ARDS. These findings suggest that earlier treatment for patients who develop more severe forms of COVID-19 may prevent unwanted outcomes. Secondly, there is additional evidence that remdesivir can speed recovery and reduce hospital days among patients with COVID-19. Finally, there is promising data that simple changes in ED care and hospital practices may improve outcomes. For example, "awake proning," which involves positioning an awake, non-intubated patients at regular intervals onto their abdomen with their face down can enable greater recruitment of lung tissue for oxygen exchange and reduce the need for subsequent intubation and mechanical ventilation. These sorts of interventions can reduce the days that patients spend in the hospital, prevent complications such as ventilator associated pneumonia, and reduce mortality related to COVID-19.

Respiratory decline needs to be identified early for patients to benefit from early medical interventions. Respiratory decline can be (a) signaled when patients report the sensation of feeling "shortness of breath" or "difficulty breathing" (i.e., dyspnea), or (b) identified when the concentration of oxygen in patients' blood or oxygen saturation are objectively measured. Current models of care ("Usual Care"), even with expanded telemedicine access, rely on patients contacting providers - a reactive process. This reactive process can delay care because most primary care practices use an intermediary (e.g., a staff member or message inbox) to screen communications for busy clinicians. Many practices do not respond to patients' concerns efficiently overnight or on weekends. These processes frustrate patients because they are concerned about contacting their providers for mild changes, irrespective of the time or day the event is occurring, because they are concerned about respiratory failure. This process is even harder for patients with limited primary care or telemedicine access or language barriers, problems disproportionately faced by Black and Latino communities. In contrast, COVID Watch is a proactive process, requesting patients report symptoms twice a day, and patients can trigger a phone call to a nurse within an hour by simply texting. COVID Watch + pulse oximetry mirrors COVID Watch but can proactively detect respiratory decline using an objective measure of oxygen saturation. In addition, COVID Watch is available free of charge and is now available in Spanish, with over 85 Spanish speaking patients enrolled to date.

To not overburden emergency departments (EDs), respiratory decline needs to be identified accurately. Both unnecessary escalations of care to the ED for patients with mild COVID-19 and delayed detection of respiratory decline in patients with severe COVID-19 may occur when managing patients with COVID-19. For usual care and COVID Watch, clinicians are reliant on the subjective sensation of dyspnea. Dyspnea is concerning enough that patients are often redirected to an urgent care center or emergency department so patients can have their oxygen saturation measured. Referring patients with an oxygen saturation <94% would justify redirecting patients to the ED for additional clinical evaluation and supportive therapy. Referring patients with mild dyspnea who turn out to have a normal oxygen saturation may be a burden to patients and their families and requires additional resource from EDs and hospitals. During times of rapid rises in community infection rates, or surges, efficient resource allocations are imperative for supporting patients who are critically ill. At the same time, patients still benefit from enhanced connections with clinical providers to reassure them that they are not experiencing respiratory decline. COVID Watch, supplemented by pulse oximetry, could provide this highly responsive team of clinicians objective data so they can accurately assess a patient's respiratory state.

In an alternative scenario, patients may have low oxygen saturation without the sensation of dyspnea, a phenomenon unique to COVID-19 infected patients, and is commonly known as "silent" or "happy" hypoxemia. These patients receive medical interventions late because they are unaware they are hypoxemic. There have been reports of COVID-19 patients arriving in EDs with profoundly low oxygen saturation levels with relatively little or no dyspnea. This has led to proposals to use home pulse oximetry to detect silent hypoxemia which have been widely reported in the media (e.g. New York Times) and resuscitation medicine forums. To address this phenomenon, the Vermont Department of Public Health has implemented a program to mail pulse oximeters to newly diagnosed COVID-19 cases 24-48 hours after contact tracing interviews. But as reported in Science: "No one, however, has studied whether early detection of hypoxia might head off bad outcomes. Some physicians believe pulse oximeters are best used with a doctor's guidance, perhaps through telemedicine. With many COVID-19 patients frightened to visit a hospital and arriving only when their symptoms have dangerously advanced, doctors also wonder whether home monitoring could hasten treatment-and whether, for some, that could make all the difference."

Based on lack of studies determining whether pulse oximetry can hasten treatment for patients deteriorating at home relative to the current standard of care in the health system of automated text messaging paired with telemedicine, the investigators believe there is equipoise between these two treatment strategies: automated text messaging with telemedicine vs. automated text messaging with telemedicine plus pulse oximetry. Therefore, a randomized comparison is needed to guide health system programs to better address this pandemic.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected or confirmed COVID-19 started on COVID Watch as routine care via (1) outpatient COVID-19 testing or (2) who were tested for COVID-19 and discharged from the ED.

Exclusion Criteria:

* less than 18 years of age
* were provided a pulse oximeter upon discharge from the ED (available for distribution as usual care for patients with suspected COVID-19 being discharged from the ED with an ED pulse ox less than 95%, who have an infiltrate on chest x-ray, are greater than 60 years of age, or who are deemed by the ED clinician to have significant comorbid conditions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2097 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- COVID Watch + Pulse Oximeter: This arm is COVID Watch + pulse oximeter device. Patients sent a pulse oximeter will be prompted twice daily to text their oxygen saturation level after walking in place for 1 minute. If the oxygen saturation is >3% lower than than the baseline first O2 sat measurement, or if it falls below an absolute level of 90%, the patient will receive an immediate call from the same on-call RN's for COVID Watch and undergo the same triage protocol .
  pulse oximeter: Patients will be prompted twice daily to text their oxygen saturation level after walking in place for 1 minute. If the oxygen saturation is >3% lower than than the baseline first O2 sat measurement, or if it falls below an absolute level of 90%, the patient will receive an immediate call from the same on-call RN's for COVID Watch and undergo the same triage protocol .
  COVID Watch: Enrolled patients receive text-based assessments, two times a day for 14 days and escalates care to a nurse via telemedicine for any reported worsening of symptoms not severe enough to recommend going to the ED immediately.
Period: Overall Study
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Started | 1041 | 1056
Completed | 1024 | 1025
Not Completed | 17 | 31
Not completed — Patients in alternate home program (e.g., home health care, inpatient rehab, etc.) were unenrolled. | 17 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter | Total
Number analyzed (Participants) | 1024 | 1025 | 2049
Age, Customized [Count of Participants; unit: Participants] — n (%)
  Participants
    <40 yo | 35 | 364 | 399
    40-49 yo | 173 | 156 | 329
    50-59 yo | 198 | 229 | 427
    60-69 yo | 179 | 161 | 340
    70 or older | 116 | 115 | 231
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 611 | 607 | 1218
  Male | 413 | 418 | 831
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 63 | 75 | 138
  Non-Hispanic Black | 347 | 350 | 697
  Non-Hispanic White | 499 | 495 | 994
  Other/Unknown | 115 | 105 | 220
Pre-Existing Conditions, n (%) [Count of Participants; unit: Participants]
  Hypertension | 334 | 329 | 663
  Diabetes | 156 | 159 | 315
  Hyperlipidemia | 247 | 259 | 506
  Chronic heart failure | 25 | 26 | 51
  Atrial fibrillation | 37 | 44 | 81
  Cancer | 103 | 109 | 212
  Chronic obstructive pulmonary disease | 29 | 34 | 63
  Asthma | 123 | 130 | 253
  Venous thromboembolism | 29 | 42 | 71
  Chronic kidney disease | 51 | 50 | 101
  History of transplant | 31 | 39 | 70
  History of substance use | 15 | 12 | 27
Insurance Coverage, n (%) [Count of Participants; unit: Participants]
  Blue Cross, Blue Shield, Commercial, or Managed Care | 340 | 302 | 642
  Medicaid or Managed Medicaid | 125 | 108 | 233
  Medicare or Managed Medicare | 137 | 137 | 274
  Other | 422 | 422 | 844

OUTCOME MEASURES:

1. Primary Outcome: Difference in Days Alive and Out of Hospital
Description: Primary outcome will be reported for patients who are confirmed to be COVID positive. Outcomes include time-based and categorical clinical outcomes. Time-based measures will be assessed at 30 days and begin when a COVID-19 patient was tested (e.g., nasopharyngeal swab) in outpatient and ED settings, or starting at the time of discharge from the hospital if enrolled in COVID Watch as an inpatient. Staying safe and out of the hospital using Days Alive and Out of Hospital (DAOH) since the date of the positive COVID-19 test. Initial analyses will include in-hospital deaths. Deaths that occur outside the hospital in 2020 will be added to a follow up analysis when National Death Index (NDI) becomes available (est. January 2021)."
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
days | 29.5 (2.3) | 29.4 (2.8)

2. Other Pre Specified Outcome: Days Alive and Out of Hospital (DAOH) by Racial/Ethnic Subgroups Among COVID-19 Positive Patients
Description: The mean number of days is per person. This data includes patients who presented to a health system hospital or any of 53 hospitals outside the health system captured in the regional health information exchange.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Groups:
- COVID Positive Black Patients - Control: Black patients enrolled in the Control arm who had a positive COVID-19 diagnosis.
- COVID Positive Hispanic Patients - Control: Hispanic patients enrolled in the Control arm who had a positive COVID-19 diagnosis.
- COVID Positive White Patients - Control: White patients enrolled in the Control arm who had a positive COVID-19 diagnosis.
- COVID Positive Other/Unknown Patients - Control: Other/Unknown (Asian, etc.) patients enrolled in the Control arm who had a positive COVID-19 diagnosis.
- COVID Positive Black Patients - Intervention: Black patients enrolled in the Intervention arm who had a positive COVID-19 diagnosis.
- COVID Positive White Patients - Intervention: White patients enrolled in the Intervention arm who had a positive COVID-19 diagnosis.
- COVID Positive Hispanic Patients - Intervention: Hispanic patients enrolled in the Intervention arm who had a positive COVID-19 diagnosis.
- COVID Positive Other/Unknown Patients - Intervention: Other/Unknown patients enrolled in the Intervention arm who had a positive COVID-19 diagnosis.
Arm/Group | COVID Positive Black Patients - Control | COVID Positive Hispanic Patients - Control | COVID Positive White Patients - Control | COVID Positive Other/Unknown Patients - Control | COVID Positive Black Patients - Intervention | COVID Positive White Patients - Intervention | COVID Positive Hispanic Patients - Intervention | COVID Positive Other/Unknown Patients - Intervention
Number analyzed (Participants) | 240 | 41 | 262 | 63 | 253 | 251 | 46 | 61
Days | 29.3 (2.6) | 29.4 (1.5) | 29.6 (2.4) | 29.6 (1.5) | 29.5 (.4) | 29.3 (3.0) | 29.1 (4.0) | 29.3 (3.0)

3. Other Pre Specified Outcome: Self-reported Anxiety Among COVID-19 Positive Patients
Description: Patients were asked to rate their anxiety (1=very worried to 5=not at all worried) on Day 0, 7, and 14.
Time Frame: 0, 7, and 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
score on a scale
  0 days | 2.9 (1.3) | 2.8 (1.3)
  7 days | 2.3 (1.3) | 2.3 (1.3)
  14 days | 2.0 (1.2) | 2.0 (1.3)

4. Other Pre Specified Outcome: Self-perception of Confidence in Managing Illness Among COVID-19 Positive Patients
Description: Patients were asked to rate their confidence that they could manage their symptoms at home (1=not at all confident to 5=very confident) on Day 0, 7, and 14.
Time Frame: 0, 7, and 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
score on a scale
  Day 0 | 4.3 (1.0) | 4.3 (1.0)
  Day 7 | 4.4 (0.9) | 4.5 (0.8)
  Day 14 | 4.5 (0.9) | 4.5 (0.8)

5. Other Pre Specified Outcome: Self-perception of Program Helpfulness in Managing Illness Among COVID-19 Positive Patients
Description: Patients were asked to rate how helpful these found the program (1=not at all helpful to 5=very helpful) on Day 0, 7, and 14.
Time Frame: 0, 7, and 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
score on a scale
  Day 0 | 4.2 (1.1) | 4.3 (1.0)
  Day 7 | 4.4 (1.0) | 4.1 (1.2)
  Day 14 | 4.6 (0.8) | 4.3 (1.1)

6. Other Pre Specified Outcome: Mortality Among COVID-19 Positive Patients
Description: The count of participants encompasses all deaths in each arm. This data includes patients who presented to a health system hospital or any of 53 hospitals outside the health system captured in the regional health information exchange.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
Participants | 3 | 5

7. Other Pre Specified Outcome: Mortality by Racial/Ethnic Subgroups Among COVID-19 Positive Patients
Description: The count of participants encompasses all deaths with respect to each arm and each race/ethnic group. This data includes patients who presented to a health system hospital or any of 53 hospitals outside the health system captured in the regional health information exchange.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | COVID Positive Black Patients - Control | COVID Positive Hispanic Patients - Control | COVID Positive White Patients - Control | COVID Positive Other/Unknown Patients - Control | COVID Positive Black Patients - Intervention | COVID Positive White Patients - Intervention | COVID Positive Hispanic Patients - Intervention | COVID Positive Other/Unknown Patients - Intervention
Number analyzed (Participants) | 240 | 41 | 262 | 63 | 253 | 251 | 46 | 61
Participants | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 2

8. Other Pre Specified Outcome: Health Care Utilization (Outpatient, Emergency Department, and Inpatient Care)
Description: The mean number of visits/hospitalizations is per patient. Emergency and Hospitalizations include patients who presented to a health system hospital or any of 53 hospitals outside the health system captured in the regional health information exchange. Office visits are within the Penn health system and do not include patients who presented to any of 53 hospitals outside the Penn health system captured in the regional health information exchange.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Number of Visits/Hospitalizations
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
Number of Visits/Hospitalizations
  ED Visits | 0.1 (0.4) | 0.1 (0.3)
  Hospitalizations | 0.1 (0.3) | 0.1 (0.3)
  Office Visits within the Health System | 0.2 (0.6) | 0.2 (0.6)

9. Other Pre Specified Outcome: Health Care Utilization (Outpatient, Emergency Department, and Inpatient Care) by Racial/Ethnic Subgroups Among COVID-19 Positive Patients
Description: The mean number of visits/hospitalizations is per patient. This data includes patients who presented to a health system hospital or any of 53 hospitals outside the health system captured in the regional health information exchange. Office visits are within the Penn health system and do not include patients who presented to any of 53 hospitals outside the Penn health system captured in the regional health information exchange.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Number of Visits/Hospitalizations
Arm/Group | COVID Positive Black Patients - Control | COVID Positive Hispanic Patients - Control | COVID Positive White Patients - Control | COVID Positive Other/Unknown Patients - Control | COVID Positive Black Patients - Intervention | COVID Positive White Patients - Intervention | COVID Positive Hispanic Patients - Intervention | COVID Positive Other/Unknown Patients - Intervention
Number analyzed (Participants) | 240 | 41 | 262 | 63 | 253 | 251 | 46 | 61
Number of Visits/Hospitalizations
  ED Visits | 0.1 (0.5) | 0.1 (0.4) | 0.1 (0.3) | 0.0 (0.2) | 0.1 (0.3) | 0.0 (0.2) | 0.1 (0.3) | 0.0 (0.2)
  Hospitalizations | 0.1 (0.4) | 0.1 (0.3) | 0.1 (0.2) | 0.1 (0.3) | 0.1 (0.3) | 0.1 (0.3) | 0.1 (0.3) | 0.1 (0.3)
  Outpatient Office Visits | 0.2 (0.4) | 0.1 (0.3) | 0.2 (0.6) | 0.1 (0.4) | 0.2 (0.4) | 0.2 (0.6) | 0.1 (0.6) | 0.2 (0.4)

10. Other Pre Specified Outcome: Incidence of Remote Monitoring Escalations to Clinician
Description: Escalations to a clinician represents the number of unique patients who escalated to a clinician one or more times throughout enrollment per their allocated study.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
Participants | 108 | 242

11. Other Pre Specified Outcome: Timing of Remote Monitoring Escalations to Clinician
Description: Mean represents average clinician response time in minutes to escalations.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
minutes | 29.7 (34.0) | 27.8 (40.5)

12. Other Pre Specified Outcome: Self-Reported Symptom Self-Management Among COVID-19 Positive Patients
Description: Patients were asked after an escalation to a clinician how they would have self-managed their COVID symptoms if not for the COVID Watch program (A. Gone to ER, B. Contacted my doctor, C. Stayed at home, or D. Other).
Time Frame: 30 days
Population: A single participant could be escalated multiple times.
Measure: Count of Units; unit: Escalations
Units Other Than Participants: Escalations
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 108 | 242
Number analyzed (Escalations) | 172 | 366
Escalations
  "Gone to the ER" | 28 | 49
  "Contacted my doctor" | 43 | 111
  "Stayed at home" | 24 | 68
  "Other" | 1 | 18
  Missing Responses | 76 | 120

13. Other Pre Specified Outcome: Days Between Program Enrollment and Home Pulse Oximetry Initiation
Description: SpO2 denotes peripheral capillary oxygen saturation. This is the number of days between when patients were enrolled to when they initiated the pulse oximetry. This only applies to the COVID Watch + Pulse Oximeter patients.
Time Frame: 30 days
Population: The control arm was not given pulse oximeters for SpO2 to be measured as per study design.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1025
Days | 2.4 (2.4)

14. Other Pre Specified Outcome: Timing of Initial Presentation of Covid-19 Positive Patients Who Returned to Emergency Department
Description: Days from enrollment to ED return visit includes patients who presented to any of 53 hospitals outside the health system captured in the regional health information exchange. ED denotes Emergency Department. Days from enrollment to ED return visit in Penn Health System does not include patients who presented to any of 53 hospitals outside the health system captured in the regional health information exchange. ED denotes Emergency Department.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
Days
  Days from enrollment to ED return visit | 10.0 (7.5) | 9.1 (7.1)
  Days from enrollment to ED return visit in Penn Health System | 10.1 (7.5) | 9.0 (7.2)

15. Other Pre Specified Outcome: Severity of Initial Presentation of Covid-19 Positive Patients Who Returned to Emergency Department as Measured by Oxygen Saturation
Description: Lowest recorded oxygen saturation percentage does not include patients who presented to any of 53 hospitals outside the health system captured in the regional health information exchange. ED denotes Emergency Department.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Oxygen Saturation (%)
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
Oxygen Saturation (%) | 96.9 (1.9) | 94.9 (4.9)

16. Other Pre Specified Outcome: Incidence of Subsequent Emergency Department Referrals
Description: Total escalations represent number of total escalations, including multiple from same patient. Clinical recommendations, including referrals, followed an pre-specified clinical protocol
Time Frame: 30 days
Measure: Number; unit: referrals
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
Number analyzed (Participants) | 1024 | 1025
referrals | 10 | 13

ADVERSE EVENTS:
Time Frame: 2 months, 1 week.
Arm/Group | COVID Watch | COVID Watch + Pulse Oximeter
All-Cause Mortality (participants affected / at risk) | 3/1024 | 5/1025
Serious Adverse Events (participants affected / at risk) | 0/1024 | 0/1025
Other Adverse Events (participants affected / at risk) | 0/1024 | 0/1025

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT04581863/Prot_SAP_000.pdf